CLINICAL TRIAL: NCT01502319
Title: Military Suicide Research Consortium
Acronym: MSRC
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: COMIRB 11-0304
Record Dates: First submitted 2011-12-09; First posted 2011-12-30 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Suicidal and Self-injurious Behaviour
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All subjects: Group/Cohort label is not applicable to this umbrella protocol. The Consortium funds specific research teams who will determine the number of group(s)/cohort(s) relevant to their study.
  Interventions: Behavioral: Cognitive therapy

INTERVENTIONS:
Behavioral: Cognitive therapy — Interventional studies conducted by the consortium focus on a range of cognitive and cognitive-behavioral techniques including cognitive therapy.

SUMMARY:
The Consortium's overall mission can be summarized as follows; each function is developed with the goal of clear military relevance:

1. Produce new scientific knowledge about suicidal behavior in the military that improves mental health outcomes for the investigators men and women in uniform.
2. Use high quality research methods and analyses to address problems in policy and practice that have a direct impact on suicide-related and other mental health outcomes for military personnel.
3. Disseminate Consortium knowledge, information, and findings through a variety of methods appropriate for decision makers, practitioners, and others who are accountable for ensuring the mental health of military personnel. This includes the rapid response function so that queries from decision makers and others to the Consortium are answered with speed and efficiency. Technical assistance and support for decision makers and others is an integral aspect of this Consortium function. This aspect of the Consortium will warehouse knowledge about suicidal behavior in general (e.g., from civilian and international sources as well as from military sources), so that military issues can be informed in a comprehensive manner.
4. Train future leaders in military suicide research through experience within a multi-disciplinary setting for Ph.D. students and postdoctoral scholars interested in research questions on military suicide of both a basic and applied nature.

DETAILED DESCRIPTION:
This is a research consortium responsible for the conduct of a wide range of studies, including clinical trials. All clinical trials funded through the consortium will be registered separately.

ELIGIBILITY:
Inclusion Criteria:

* MSRC studies are inclusive of all individuals who are eligible as defined by each study's protocol regardless of age, gender, race or ethnicity, socioeconomic status, sexual orientation, and any other demographic characteristics. Measures and treatments are translated and culturally adapted to the extent possible.

Exclusion Criteria:

* Specific to each investigator's protocol.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Given the age range of active duty military, reservists, and veterans, it is expected that funded Study Principal Investigators will enroll subjects that are young adults (18 to 21 years) to Senior Citizens (over 65 years).
Sampling Method: Probability Sample
Enrollment: 5400 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Suicide | varies by study
  Specific outcomes related to suicide will vary as a function of the individual studies conducted within the consortium

SECONDARY OUTCOMES:
Suicide | varies by study
  Secondary outcomes related to suicide will vary as a function of the individual studies conducted within the consortium.

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Gutierrez, PhD, Principal Investigator — VA Eastern Colorado Health Care System
Locations (1):
- Denver VA Medical Center, Denver, Colorado, United States

REFERENCES:
- See also: Consortium website, click here for more information — http://msrc.fsu.edu/
- See also: Principal investigator organization website, click here for more information — http://www.mirecc.va.gov/visn19/